CLINICAL TRIAL: NCT00641862
Title: Randomized Trial of Vitamin B12 in Pregnant Indian Women
Acronym: B12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: St. John's Research Institute (Other)
Responsible Party: Principal Investigator, Christopher Duggan, Professor in the Department of Nutrition, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HD052143
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Pregnancy
Keywords: Pregnancy; Maternal Nutritional Status; Vitamin B12
MeSH Terms: interventions — Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin B12 (Active Comparator): Vitamin B12
  Interventions: Dietary Supplement: Vitamin B12
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin B12 — Daily oral administration of 50 µg of Vitamin B12 taken from enrollment (at or before 14 weeks gestational age) until delivery
  Arms: Vitamin B12
Other: Placebo — Placebo taken daily from enrollment (at or before 14 weeks gestational age) until delivery
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind trial among 300 pregnant Indian women in order to determine the effectiveness of vitamin B12 supplementation in improving maternal B12 status. Secondary aims for this trial include maternal hemoglobin, maternal weight gain during pregnancy and infant birthweight. All women will receive standard of prenatal obstetric care, including routine supplementation with iron and folate.

DETAILED DESCRIPTION:
The incidence of poor fetal growth and adverse maternal and infant birth outcomes is quite high in India, and several lines of evidence suggest that maternal nutritional status may be an important factor. We have previously performed extensive evaluations of poor fetal and infant outcomes in other settings, and found that maternal micronutrient supplementation (B vitamins including vitamin B12, plus vitamins C and E) in HIV positive Tanzanian mothers decreased the risk of low birthweight (<2500 g) by 44% (RR (95% CI) 0.56 (0.38-0.82)), severe preterm birth (<34 weeks of gestation) by 39% (RR 0.61 (0.38-0.96)), and small size for gestational age at birth by 43% (RR 0.57 (0.39-0.82)). In a prospective cohort study of 410 pregnant Indian women, we recently found a strong relationship between maternal serum vitamin B12 concentration and risk of infant intrauterine growth retardation (IUGR). Compared to women in the highest tertile of serum B12 concentration, women in the lowest tertile were significantly more likely to have IUGR infants, after controlling for maternal age, weight, education, and parity (OR (95% CI) 5.98 (1.72-20.74)). We now propose a randomized, double-blind trial among 300 pregnant Indian women in order to determine the effectiveness of vitamin B12 supplementation (50 µg daily) in improving maternal B12 status. Secondary aims for this exploratory trial include maternal hemoglobin, maternal weight gain during pregnancy and infant birthweight. All women will receive standard of prenatal obstetric care, including routine supplementation with iron and folate. The study will be a collaborative effort between the Division of Nutrition, St John's Research Institute, Bangalore, India, and the Department of Nutrition, Harvard School of Public Health, Boston, US.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at or before 14 weeks gestational age.

Exclusion Criteria:

* Women who anticipate moving outside of the study area before study completion
* Those with twin or multiple pregnancies
* Those who test positive for hepatitis B (HepBSAg), HIV or Syphilis (VDRL)
* Those taking vitamin supplements in addition to folate and iron
* Those with a serious pre-existing medical condition, defined as conditions that require chronic or daily medical therapy such as connective tissue diseases, hypertension not related to pregnancy, inflammatory bowel disease, active tuberculosis, symptomatic heart disease, and insulin dependent diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2008-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Duggan, MD, MPH, Principal Investigator — Harvard School of Public Health (HSPH); Anura Kurpad, MBBS, PhD, Principal Investigator — St. John's Research Institute; Krishnamachari Srinivasan, MD, Principal Investigator — St. John's Research Institute
Locations (1):
- St. John's Medical Research Institute, St. John's National Academy of Health Sciences, Bangalore, Karnataka, India

REFERENCES:
- [Background] Muthayya S, Dwarkanath P, Mhaskar M, Mhaskar R, Thomas A, Duggan C, Fawzi WW, Bhat S, Vaz M, Kurpad A. The relationship of neonatal serum vitamin B12 status with birth weight. Asia Pac J Clin Nutr. 2006;15(4):538-43. PMID 17077072
- [Background] Muthayya S, Kurpad AV, Duggan CP, Bosch RJ, Dwarkanath P, Mhaskar A, Mhaskar R, Thomas A, Vaz M, Bhat S, Fawzi WW. Low maternal vitamin B12 status is associated with intrauterine growth retardation in urban South Indians. Eur J Clin Nutr. 2006 Jun;60(6):791-801. doi: 10.1038/sj.ejcn.1602383. Epub 2006 Jan 11. PMID 16404414
- [Derived] Finkelstein JL, Fothergill A, Venkatramanan S, Layden AJ, Williams JL, Crider KS, Qi YP. Vitamin B12 supplementation during pregnancy for maternal and child health outcomes. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD013823. doi: 10.1002/14651858.CD013823.pub2. PMID 38189492
- [Derived] Srinivasan K, Thomas S, Anand S, Jayachandra M, Thomas T, Strand TA, Kurpad AV, Duggan CP. Vitamin B-12 Supplementation during Pregnancy and Early Lactation Does Not Affect Neurophysiologic Outcomes in Children Aged 6 Years. J Nutr. 2020 Jul 1;150(7):1951-1957. doi: 10.1093/jn/nxaa123. PMID 32470975
- [Derived] Anand S, Thomas S, Jayachandra M, Thomas T, Strand TA, Kurpad AV, Duggan CP, Srinivasan K. Effects of maternal B12 supplementation on neurophysiological outcomes in children: a study protocol for an extended follow-up from a placebo randomised control trial in Bangalore, India. BMJ Open. 2019 Feb 19;9(2):e024426. doi: 10.1136/bmjopen-2018-024426. PMID 30782904
- [Derived] Winje BA, Kvestad I, Krishnamachari S, Manji K, Taneja S, Bellinger DC, Bhandari N, Bisht S, Darling AM, Duggan CP, Fawzi W, Hysing M, Kumar T, Kurpad AV, Sudfeld CR, Svensen E, Thomas S, Strand TA. Does early vitamin B12 supplementation improve neurodevelopment and cognitive function in childhood and into school age: a study protocol for extended follow-ups from randomised controlled trials in India and Tanzania. BMJ Open. 2018 Feb 22;8(2):e018962. doi: 10.1136/bmjopen-2017-018962. PMID 29472265
- [Derived] Duggan C, Srinivasan K, Thomas T, Samuel T, Rajendran R, Muthayya S, Finkelstein JL, Lukose A, Fawzi W, Allen LH, Bosch RJ, Kurpad AV. Vitamin B-12 supplementation during pregnancy and early lactation increases maternal, breast milk, and infant measures of vitamin B-12 status. J Nutr. 2014 May;144(5):758-64. doi: 10.3945/jn.113.187278. Epub 2014 Mar 5. PMID 24598885
- [Derived] Lukose A, Ramthal A, Thomas T, Bosch R, Kurpad AV, Duggan C, Srinivasan K. Nutritional factors associated with antenatal depressive symptoms in the early stage of pregnancy among urban South Indian women. Matern Child Health J. 2014 Jan;18(1):161-170. doi: 10.1007/s10995-013-1249-2. PMID 23440491

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin B12 | Placebo
Started | 183 | 183
Completed | 139 | 145
Not Completed | 44 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin B12 | Placebo | Total
Number analyzed (Participants) | 183 | 183 | 366
Age, Continuous [Median (Inter-Quartile Range); unit: years] — We confirm that the median and inter-quartile ranges listed here are correct
  years | 22 [20 to 24] | 22 [20 to 24] | 22 [20 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 183 | 366
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Maternal Serum B12 Concentration From 1st to 3rd Trimester
Time Frame: from 1st to 3rd trimester
Population: Serum samples were available for analysis among 102 of the original 183 participants in each arm.
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Vitamin B12 | Placebo
Number analyzed (Participants) | 102 | 102
pmol/L | 3.0 [-54.8 to 83.5] | -37.6 [-66.5 to -10.9]

2. Secondary Outcome: Cognitive Scale, Bayley Scales of Infant Development, 3rd Edition
Description: The cognitive scale is a single scale that measures sensorimotor integration, concept formation, attention, habituation, and memory. Higher values represent better performance. The interquartile range provides an adequate assessment of the variability of the data. The minimum possible score of the cognitive scale is 0 and the maximum possible score is 91.
Time Frame: 9 months
Population: Outcome was measured among 178 of the 366 enrolled participants.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Vitamin B12 | Placebo
Number analyzed (Participants) | 78 | 100
units on a scale | 39 [37 to 41] | 39.5 [38 to 42]

3. Secondary Outcome: Receptive Language Scale, Bayley Scales of Infant Development, 3rd Edition
Description: The Receptive Language Scale is a single scale that measures the ability of the child to recognize sounds and understand spoken words and directions. Higher values represent better performance. The interquartile range provides adequate assessment of the variability of the data. The minimum possible score is 0 and the maximum possible score is 49.
Time Frame: 9 months
Population: This outcome was measured among 178 of the 366 enrolled participants.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Vitamin B12 | Placebo
Number analyzed (Participants) | 78 | 100
units on a scale | 11 [11 to 12] | 11 [11 to 12]

4. Secondary Outcome: Expressive Language Scale, Bayley Scales of Infant Development, 3rd Edition
Description: The Expressive Language Scale is a single scale that measures the ability of the child to communicate using sounds, gestures, or words. Higher scores represent better performance. The interquartile range provides adequate assessment of the variability of the data. The minimum possible value is 0 and the maximum possible value is 48.
Time Frame: 9 months
Population: This outcome was measured in 178 of the 366 enrolled participants
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Vitamin B12 | Placebo
Number analyzed (Participants) | 78 | 100
units on a scale | 10 [9 to 12] | 11 [9 to 12]

5. Secondary Outcome: Fine Motor Scale, Bayley Scales of Infant Development, 3rd Edition
Description: The Fine Motor Scale is a single scale that measures prehension, perceptual-motor integration, motor planning and speed, visual tracking, reaching, object grasping, object manipulation, functional hand skills, and responses to tactile information. Higher values represent better performance. The interquartile range provides adequate assessment of the variability of the data. The minimum possible value is 0 and the maximum possible value is 66.
Time Frame: 9 months
Population: This outcome was measured in 178 of the original 366 participants
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Vitamin B12 | Placebo
Number analyzed (Participants) | 78 | 100
units on a scale | 26 [25 to 27] | 26 [25 to 27]

6. Secondary Outcome: Gross Motor Scale, Bayley Scales of Infant Development, 3rd Edition
Description: The Gross Motor Scale is a single scale that measures movement of the limbs and torso, static positioning (e.g., sitting, standing), dynamic movement including locomotion and coordination, balance, and motor planning. Higher values represent better performance. The interquartile range provides adequate assessment of the variability of the data. The minimum possible value is 0 and the maxiumum possible value is 72.
Time Frame: 9 months
Population: This outcome was measured in 178 of the 366 enrolled participants
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Vitamin B12 | Placebo
Number analyzed (Participants) | 78 | 100
units on a scale | 36 [31 to 38] | 34 [30 to 38]

7. Secondary Outcome: Kaufman's Assessment Battery for Children (KABC)
Description: This test is used for assessing child intelligence
Time Frame: 60-72 months
Reporting Status: Not Posted

8. Secondary Outcome: The Wechsler Preschool and Primary Scale of Intelligence (WPPSI)
Description: WPPSI is an intelligence test designed for children ages 2 years 6 months to 7 years 7 months. It is a paper-pencil test that will be administered during the 78 month follow up to assess child's intellectual functioning.
Time Frame: 78 months
Reporting Status: Not Posted

9. Secondary Outcome: Vineland Social Maturity Scale (VSMS)
Description: This scale has 8 main domains which include, Self Help General, Self Help Dressing, Self Direction, Occupation, Communication, Locomotion and Socialization. It is possible to calculate Social age and Social quotient from VSMS which will provide a good idea about the social maturity of the infant. VSMS will be used in conjunction with KABC at age 60-72 months of age.
Time Frame: 60-72 months
Reporting Status: Not Posted

10. Secondary Outcome: The Brief P Test
Description: The Brief P test is a measure of infant executive function based on parental rating. It will be administered at 66 months postpartum.
Time Frame: 66 months postpartum
Reporting Status: Not Posted

11. Secondary Outcome: Parental Version of Strengths and Difficulties Questionnaire (SDQ)
Description: Administered at 78 months to assess childhood behavioral problems. The SDQ has 25 items and generates 5 scales: emotional problem, conduct problem, hyperactivity/inattention, peer relationship problems and pro-social behavior.
Time Frame: 78 months
Reporting Status: Not Posted

12. Secondary Outcome: Bradley Infant-Toddler Home Tools
Description: Home tools used to analyze aspects of home environment. This scale captures information on parenting behavior under 6 domains: responsivity, acceptance, organization, learning materials, parental involvement, and variety of stimulation at home). Trained study personnel will administer this questionnaire to participating families at 60 months.
Time Frame: 60 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Vitamin B12 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/183 | 0/183
Other Adverse Events (participants affected / at risk) | 0/183 | 0/183

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No